CLINICAL TRIAL: NCT02654093
Title: A Randomized, Open-label, Single-dose, 3-period, 6-sequence Crossover Study to Evaluate the Safety and the Pharmacokinetics After Oral Concurrent Administration of Raloxifene, Cholecalciferol in Healthy Korean Male Subjects
Brief Title: A Drug-drug Interaction Study of DP-R213
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DP-CTR213-I-02
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — Cholecalciferol; Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A (Experimental): A → B → C / A: Cholecalciferol, B: Raloxifene, C: Cholecalciferol+Raloxifene
  Interventions: Drug: Cholecalciferol; Drug: Raloxifene; Drug: Cholecalciferol and Raloxifene co-administration
- Group B (Experimental): A → C → B
  Interventions: Drug: Cholecalciferol; Drug: Raloxifene; Drug: Cholecalciferol and Raloxifene co-administration
- Group C (Experimental): B → A → C
  Interventions: Drug: Cholecalciferol; Drug: Raloxifene; Drug: Cholecalciferol and Raloxifene co-administration
- Group D (Experimental): B → C → A
  Interventions: Drug: Cholecalciferol; Drug: Raloxifene; Drug: Cholecalciferol and Raloxifene co-administration
- Group E (Experimental): C → A → B
  Interventions: Drug: Cholecalciferol; Drug: Raloxifene; Drug: Cholecalciferol and Raloxifene co-administration
- Group F (Experimental): C → B → A
  Interventions: Drug: Cholecalciferol; Drug: Raloxifene; Drug: Cholecalciferol and Raloxifene co-administration

INTERVENTIONS:
Drug: Cholecalciferol
Drug: Raloxifene
Drug: Cholecalciferol and Raloxifene co-administration

SUMMARY:
The purpose of this study is to learn about the effect of raloxifene on how the body absorbs and processes cholecalciferol and how cholecalciferol affects raloxifene when they are taken together.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age above 19
* The result of Ideal Body Weight(IBW) is not less than -20%, no more than +20%
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial.

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment in completion of this clinical study
* Treatment history of other drugs within last 10 days

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve(AUCt) of raloxifene | 0, 2, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96 hours
Peak plasma concentration(Cmax) of raloxifene | 0, 2, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96 hours
AUCt,corr of cholecalciferol | -20, -16, -12, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 84 hours
Cmax,corr of cholecalciferol | -20, -16, -12, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 84 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungbook National University Hospital, Jung-gu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HW, Kang WY, Jung W, Gwon MR, Cho K, Lee B, Seong SJ, Yoon YR. Pharmacokinetic Drug Interaction Between Raloxifene and Cholecalciferol in Healthy Volunteers. Clin Pharmacol Drug Dev. 2022 May;11(5):623-631. doi: 10.1002/cpdd.1062. Epub 2022 Jan 4. PMID 34984851